CLINICAL TRIAL: NCT06825182
Title: Survey on the Current Status of Islet Alpha Cell Function in Patients with Type 2 Diabetes and Interventional Study of GLP-1RA: a Multicenter, Prospective Study
Brief Title: Current Status of Islet Alpha Cell Function in Patients with Type 2 Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20240514-11
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Islet Alpha Cell Function; Glucagon-Like Peptide-1 Receptor Agonists (GLP1-RA)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Loxenatide (Other)
  Interventions: Drug: Outpatient newly diagnosed type 2 diabetes subjects; Drug: Inpatient newly diagnosed type 2 diabetes subjects

INTERVENTIONS:
Drug: Outpatient newly diagnosed type 2 diabetes subjects — Outpatient newly diagnosed type 2 diabetes subjects, who have signed the informed consent form, meet the inclusion and exclusion criteria, and have their demographic data collected, including height, weight, systolic and diastolic blood pressure, and calculation of the body mass index (BMI) = weight/height^2 (kg/m^2). Fasting and postprandial 120-minute glucose, insulin (INS), C-peptide (Cp), and glucagon (GCG) levels are measured, or an Oral Glucose Tolerance Test (OGTT) is performed, measuring glucose, INS, Cp, GCG at 0, 30, and 120 minutes, and renal function and HbA1c are tested, with eGFR calculated. Type 2 diabetes patients are treated with GLP-1RA for three months, and then the aforementioned indicators are retested to complete the study.
Drug: Inpatient newly diagnosed type 2 diabetes subjects — Demographic data are collected. Fasting and postprandial 120-minute glucose, insulin (INS), C-peptide (Cp), and glucagon (GCG) levels are measured, or an Oral Glucose Tolerance Test (OGTT) is conducted, measuring glucose, INS, Cp, GCG at 0, 30, and 120 minutes, and renal function and HbA1c are tested. During hospitalization, if hypoglycemic symptoms occur or peripheral blood glucose or continuous glucose monitoring is ≤3.9 mmol/L, immediate venous blood is drawn for glucose, GCG, adrenocorticotropic hormone (ACTH), cortisol (Cor), growth hormone (GH), and Cp testing. Patients are treated with GLP-1RA for three months, then the aforementioned indicators are retested to complete the study and hypoglycemia (including hypoglycemic clamp and hypoglycemia tests) is assessed for glucose and GCG, with additional tests for ACTH, Cor, GH, and Cp if conditions permit, to complete the study.

SUMMARY:
By detecting the fasting and postprandial 120-minute glucose, insulin (Insulin, INS), C-peptide (C-peptide, Cp), glucagon (GCG) levels in newly diagnosed type 2 diabetes patients, or the 0-minute, 30-minute, 120-minute glucose, INS, Cp, GCG levels during the Oral Glucose Tolerance Test (OGTT), and examining the glucose, INS, Cp, GCG levels during hypoglycemia, the current status of islet alpha cell function in diabetic patients is observed. Type 2 diabetes patients willing to participate are treated with GLP-1RA for 3 months, and then retested for fasting and postprandial 120-minute glucose, INS, Cp, GCG, or the 0-minute, 30-minute, 120-minute glucose, INS, Cp, GCG during OGTT, as well as the counter-regulatory hormone levels during hypoglycemia, to assess the improvement of islet alpha cell function by GLP-1RA.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate voluntarily and able to sign the Informed Consent Form before the trial;
* Newly diagnosed patients with type 2 diabetes, aged 18 years or older, meeting the WHO 1999 diagnostic criteria;
* Subjects who are capable and willing to maintain a regular diet and exercise regimen.

Exclusion Criteria:

* Patients who are allergic to GLP-1RA or have a BMI less than 24 kg/m^2;
* History of using blood sugar-lowering medications;
* Estimated glomerular filtration rate (eGFR) less than 30 ml/(min*1.73 m^2);
* History of drug abuse or alcohol dependence within the past 5 years;
* Patients with poor compliance and irregular diet and exercise;
* History of diagnosed pancreatitis, pancreatic tumor, medullary thyroid carcinoma, or diabetic retinopathy stage IV or higher;
* Patients who have used systemic glucocorticoid therapy within the past 3 months;
* Presence of infection or stress within the past four weeks;
* Any other significant condition or comorbidity judged by the researcher, such as severe cardiopulmonary disease, endocrine disorders, neurological disorders, tumors, other pancreatic diseases, mental illness, history of alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucagon levels | 19 months
  Compare the glucagon levels in diabetic subjects during hyperglycemia and hypoglycemia, and the changes in GCG after 3 months of GLP-1RA treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hostital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No